CLINICAL TRIAL: NCT05397158
Title: Study on Optimization of Intestinal Preparation Before Colonoscopy in Older Patients
Brief Title: Optimization of Intestinal Preparation in Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: YuHe
Record Dates: First submitted 2022-05-18; First posted 2022-05-31 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2022-07

CONDITIONS: Colonoscopy; Older Adults
Keywords: colonoscopy; intestinal preparation; older adults
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Endoscopist blind method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single administration of low dose polyethylene glycol group (Experimental): The patients take 30ml lactulose in the morning 1 day before the examination, and eat without residue in lunch and dinner; Take 2L PEG in the morning of the examination day and fast at breakfast and lunch of the day.
  Interventions: Procedure: single administration of low dose polyethylene glycol
- control group (Active Comparator): The patients in control group take 2L PEG the day before the examination, fast at dinner (patients without diabetes) and eat without residue (patients with diabetes). Patients take 2L PEG again in the morning of the examination day, and fasted at breakfast and lunch of the day.
  Interventions: Procedure: single administration of low dose polyethylene glycol

INTERVENTIONS:
Procedure: single administration of low dose polyethylene glycol — Patients in single administration of low dose polyethylene glycol (PEG) group: Take 30ml lactulose and 2L PEG.
  Patients in control group: Take 4L PEG.

SUMMARY:
Older adults are susceptible to intestinal tumors. Colonoscopy can screen colorectal cancer, adenoma and other diseases. There is a large demand for colonoscopy in the older adults, and the risk during peri-colonoscopy period is high. According to the common intestinal preparation methods and the characteristics of the older adults, the investigators propose a modified method, that is single administration of low dose polyethylene glycol (PEG). Specifically, take 30ml lactulose in the morning 1 day before the examination, and eat without residue in lunch and dinner, Take 2L PEG in the morning of the examination day and fast at breakfast and lunch of the day. Taking 4L PEG in 2 days as the control group. The fasting and diarrhea period is shorter in the modified group than that in the control group, and the dose of PEG is less. Lactulose, a laxative, is taken one day before the examination, and the intestinal preparation time is longer than that of single administration. The situation of comfort, sleep and fecal incontinence during the intestinal preparation of the two groups will be compared. The results of electrolyte, blood glucose and B-type brain natriuretic peptide between the two groups will be also compared. The effect of intestinal preparation will be evaluated by the standardization of Boston intestinal preparation scale, and endoscopist blind method will be used in colonoscopy.

DETAILED DESCRIPTION:
The participants in control group take 2L PEG the day before the examination, fast at dinner (participants without diabetes) and eat without residue (participants with diabetes). Participants take 2L PEG again in the morning of the examination day, and fasted at breakfast and lunch of the day.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 50y
* Colonoscopy is planned
* Willing to participate

Exclusion Criteria:

* Age<50y
* Unwilling to participate
* Missing data

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Intestinal preparation Cleanliness assessment | Up to 1 hour
  The effect of intestinal preparation will be evaluated by Boston Intestinal Preparation Scale.The minimum score is 0，and the maximum score is 9. Higher scores mean a better outcome. Endoscopist blind method will be used.

SECONDARY OUTCOMES:
Blood potassium level before and after intestinal preparation | Up to 1 week
  Blood potassium in mmol/L.
Blood sodium level before and after intestinal preparation | Up to 1 week
  Blood sodium in mmol/L.
Blood glucose level before and after intestinal preparation | Up to 1 week
  Blood glucose in mmol/L.
B-type brain natriuretic peptide (BNP) level before and after intestinal preparation | Up to 1 week
  BNP in pg/ml.
The situation of comfort during the intestinal preparation | Two days
  Comfort situation questionnaire. The score of comfort questionnaire is 1 to 10, 1 represents extremely uncomfortable and 10 represents very comfortable.
The situation of sleep during the intestinal preparation | One day
  Sleep situation questionnaire. The length of sleep in hour, the number of awakening, the number of urination and defecation.
The situation of fecal incontinence during the intestinal preparation | One day
  Fecal incontinence questionnaire. Does the patient have fecal incontinence and the number of fecal incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No